CLINICAL TRIAL: NCT02236260
Title: Evaluation of the Benefit Provided by the Addition of Acupunctural Analgesia With Electrostimulation to Conventional Local Anesthesia Compared to Conventional Local Anesthesia Alone in Surgery of Deep Brain Stimulation for Movement Disorders.
Brief Title: Evaluation of the Benefit Provided by Acupuncture During a Surgery of Deep Brain Stimulation
Acronym: ACUplus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC14_0060
Record Dates: First submitted 2014-08-29; First posted 2014-09-10 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Electroacupuncture; Anesthesia, Local; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anesthesia alone (Active Comparator)
  Interventions: Drug: Local Anesthesia (lidocaine hydrochloride)
- Local Anesthesia + Electroacupuncture (Experimental)
  Interventions: Procedure: Electroacupuncture; Drug: Local Anesthesia (lidocaine hydrochloride)

INTERVENTIONS:
Procedure: Electroacupuncture — Acupuncture will be performed using an electrical stimulator (generating electrical stimulation) for electroacupuncture.
  Arms: Local Anesthesia + Electroacupuncture
Drug: Local Anesthesia (lidocaine hydrochloride) — All patients will receive injectable paracetamol for pain relief, a mix of nitrous oxide 50% and oxygen 50% for analgesia and lidocaine hydrochloride for local anesthesia.

SUMMARY:
The effectiveness of Deep Brain Stimulation (DBS) in certain movement disorders is widely demonstrated. The success of this procedure requires that the patient is awake and cooperative. The conditions of this intervention can be difficult to tolerate by the patient for several reasons: long procedure (from 3 to 8 hours), body immobilisation (particularly the head in the stereotactic frame), stress related to the localization of the DBS. It is therefore important to improve the comfort as well as the cooperation of the patient, during implantation of the DBS electrodes, in order to optimize the conditions of the intervention. In addition to analgesia, acupuncture should allow sedation without affecting alertness and should contribute to the regulation of any vegetative reactions during the procedure. Therefore, we hypothesize that acupuncture could improve the quality of care of the patient during a DBS procedure. In practice, this is electroacupuncture that will be used in this research to maintain the stimulation of acupuncture points to an optimal level during the time of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes aged who are >= 18 years
* Disabling movement disorders, resistant to medical treatment, in Parkinson's patients who should benefit from a Deep Brain Stimulation in the subthalamic nucleus
* Scheduled intervention of a Deep Brain Stimulation
* Understanding of acupunctural analgesia with electrostimulation
* Signed informed consent
* Membership to a social security insurance scheme

Exclusion Criteria:

* Patients who are >= 75 years
* History of intolerance to acupuncture
* Contraindications to local anesthesia
* Respiratory problems (asthma, COPD, ...)
* Holder of an implanted pacemaker
* Obesity with BMI > 30
* History of motion sickness
* Unstabilized psychiatric disorders
* Impaired cognitive functions
* Pregnancy
* Breastfeeding
* Minors
* Major under a legal protection regime

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Patient comfort, judged by "Edmonton Symptom Assessment System" scale (ESAS) | The day of the DBS procedure

SECONDARY OUTCOMES:
Patient anxiety, judged by Hamilton anxiety scale (HAMA) | The day before the DBS procedure, the day of the DBS procedure, 2 days after the DBS procedure
Drug consumption | The day of the DBS procedure, 2 days after the DBS procedure
Anesthesia monitoring parameters: heart rate, blood pressure, pulse oximetry | The day of the DBS procedure, 2 days after the DBS procedure
  Composite measure
Adverse effects | The day before the DBS procedure,the day of the DBS procedure, 2 days after the DBS procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie RAOUL, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Nantes, Nantes, France